CLINICAL TRIAL: NCT06721416
Title: Comparing the Acute Effects and Cortical Hemodynamic Response of Different Exercise Approaches in Patients With Multiple Sclerosis: fNIRS Study
Brief Title: Comparing the Acute Effects of Different Exercise Approaches in Patients With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Merve Sevik Dönderici, Principal Investigator, Acibadem University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-07/229
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; aerobic exercise; virtual reality; fatigue; cognition
MeSH Terms: conditions — Multiple Sclerosis; Fatigue

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Virtual Reality Beased (Experimental): VR based aerobic exercise
  Interventions: Other: VR Based Aerobic Exercise
- Traditional (Experimental): Cycling ergometer based aerobic exercise
  Interventions: Other: Traditional Aerobic Exercise
- Conventional (Experimental): Conventional physical therapy approaches
  Interventions: Other: Conventional Exercise

INTERVENTIONS:
Other: Traditional Aerobic Exercise — Traditional aerobic exercise will be continued with an arm ergometer, at moderate intensity, for 30 minutes.
  Arms: Traditional
Other: VR Based Aerobic Exercise — In the virtual reality-based aerobic exercise training, the game called "Beat Saber" will be played with Oculus Quest 2 virtual reality for 30 minutes.
  Arms: Virtual Reality Beased
Other: Conventional Exercise — The conventional exercise program will be modified with stabilization, balance and strengthening exercises, taking into account the functional status of the participants.
  Arms: Conventional

SUMMARY:
Multiple Sclerosis (MS) is the second most common neurological disorder in young adults after trauma. Treatments developed today can slow progression and reduce symptoms. Exercise therapy is a useful rehabilitation practice in MS to manage symptoms, restore function, optimize quality of life, ensure well-being and increase participation in daily life activities. In this study, it is planned to investigate the acute effects of conservative and virtual reality (VR)-based aerobic exercise applications and standard exercises that frequently form the rehabilitation programs of individuals with MS in clinics. For this purpose, patients with MS who met the inclusion criteria were given two-week intervals; Conservative aerobic exercise, virtual reality-based aerobic exercise and standard exercise practices will be performed. With the data obtained from this study, it is aimed to investigate the safety of aerobic exercises performed using VR tools that can be used in telerehabilitation applications, which are thought to have a very important place in MS rehabilitation in the future, in terms of acute body temperature increase, cognitive and physical fatigue caused by conservative methods and fNIRS cortical effects of VR-based aerobic exercise applications. It will be possible to prove it with objective methods such as.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as Relapsing Remitting MS by neurologist according to the McDonald Criteria.
* 18-55 years old.
* EDSS score < 4.5
* Mini mental examination test score ≥ 24
* No MS attack in the last 6 months.
* No visual or vestibular deficits.
* Signed the written consent form.

Exclusion Criteria:

* Having previous full immersive VR experience.
* Having an additional neurological disease.
* Spasticity in any muscle of the upper extremity > 3, according to MAS.
* Continuing the active physical therapy and rehabilitation program.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
Energy Spent | For 30 minutes during the entire exercise
  Sense Wear Pro3 Armband by Body Media Inc. (USA): It will be used to calculate the energy spent during exercises. This device is a 2-axis monitor with multiple sensors such as a galvanic skin response sensor to evaluate skin electrical resistance changes and a skin temperature sensor to evaluate temperature changes. The device will be worn on the individuals' right arm triceps muscle throughout the exercises and will be used to calculate the energy spent during the exercises.
Cortical Activity | During preintervention cognitive tasks, for 30 minutes during the entire exercise, during postintervention cognitive tasks
  Functional Near Infrared Light Spectroscopy (fNIRS): fNIRS is an optical system that uses near-infrared (NIR) light in the assessment of brain activity by measuring light absorption differences in changes in oxy-hemoglobin and deoxy-hemoglobin concentrations. The modified Beer-Lambert law is used to convert and calculate light intensity measurements obtained from the brain into hemodynamic changes. Hemodynamic responses that occur with different stimuli in the prefrontal cortex region of the brain can be monitored with these optical systems. In this study, it is planned to measure individuals' prefrontal cortex activations while performing 3 different exercises and a post-exercise cognitive performance test.
Body Temperature | immediately before the exercise, immediately after the exercise
  Individuals' body temperatures will be measured with the help of an electronic digital thermometer before and after the exercises.
Electrodermal Activity | During preintervention cognitive tasks, for 30 minutes during the entire exercise, during postintervention cognitive tasks
  Electrodermal activity data will be recorded with the Shimmer device to be used to determine the stress levels of the patients.
Cognitive Function | Immediately before the exercise, immediately after the exercise
  Stroop test will be used to compare the cognitive performances of the patients before and after exercise and to comment on cognitive fatigue after exercise.
Cognitive Function | Immediately before the exercise, immediately after the exercise
  2-back test will be used to compare the cognitive performances of the patients before and after exercise and to comment on cognitive fatigue after exercise.
Cognitive Function | Immediately after the exercise
  Symbol Digit Modalities Test will be used after the exercise to evaluate cognitive performance.
Physical Fatigue | Immediately after the exercise
  Modified Borg Scale will be used after the exercise to evaluate subjective physical fatigue. The values of this scale range from 0 to 10. While 0 means I have no fatigue, 10 indicates the most severe fatigue.
Satisfaction Level satisfaction level Satisfaction Level | Immediately after the exercise
  It will be evaluated with the Satisfaction Evaluation Survey of Virtual Rehabilitation Systems. The total score range in this survey varies between 6-30, with higher scores being associated with higher satisfaction.
Late-term fatigue | 24 hours later after the exercise
  One day after the exercises, patients will be questioned by phone about whether they have arm pain, and in case of pain, they will be asked to score the severity of pain according to Modified Borg Scale. The values of this scale range from 0 to 10. While 0 means I have no fatigue, 10 indicates the most severe fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Sevik Dönderici, MSc, Principal Investigator — Acibadem University
Locations (1):
- Acibadem University, Ataşehir, Istanbul, Turkey (Türkiye)